CLINICAL TRIAL: NCT07257536
Title: Xinxing Eye Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025KYPJ117
Record Dates: First submitted 2025-11-18; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Refractive Errors; Cataract
MeSH Terms: conditions — Refractive Errors; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To establish the baseline levels and monitor the progress of two newly introduced global eye health indicators in Xinxing County, including effective refractive error coverage (eREC) and effective cataract surgery coverage (eCSC). And to assess the prevalence and treatment status of common eye disease in Xinxing County.

ELIGIBILITY:
Inclusion Criteria:

* Primary and secondary school students in Xinxing County and people covered by the national basic public health service, including children aged 0-6, seniors over 65 years old and diabetic patients, etc.
* Voluntarily participate in this study and provide signed informed consent

Exclusion Criteria:

* Unable to cooperate with research-related examinations, such as those with disabilities, communication barriers, or other reasons that prevent examinations
* With serious systemic disease that may affect the examination, or participating in the research examination may endanger one's health
* Other people who the researchers consider unsuitable to participate in this study

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary and secondary school students in Xinxing County and people covered by the national basic public health service, including children aged 0-6, seniors over 65 years old and diabetic patients, etc.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | through study completion, an average of 1 year
  Test and record uncorrected visual acuity; if the participant wears glasses, measure the best corrected visual acuity with glasses. For participants with poor unaided or corrected visual acuity (<4.7), perform additional pinhole visual acuity testing.

SECONDARY OUTCOMES:
Strabismus | through study completion, an average of 1 year
  Assess strabismus status and angle at both near and distance fixation.
Autorefraction | through study completion, an average of 1 year
  Measure spherical power, cylindrical power, and axis in both eyes. Cycloplegia may be required in children, preferably using 1% tropicamide, one drop each time, three times. Before cycloplegia, check allergy history, medical history, and anterior chamber depth; inform guardians of potential risks and precautions related to cycloplegia, and ensure that guardians accompany the child throughout the procedure.
Questionnaire | through study completion, an average of 1 year
  Questionnaires on demographics, disease histories and etc.
Fundus examination | through study completion, an average of 1 year
  Examine the retina of both eyes and document any retinal pathology. If pupils are too small, mydriasis may be required, following the same drugs and procedures as above.
Anterior segment examination | through study completion, an average of 1 year
  Use a slit lamp to examine eyelids, conjunctiva, cornea, anterior chamber, and lens in both eyes. Record any abnormalities. Grade lens opacities according to the LOCS III classification system.

IPD SHARING:
Plan to Share IPD: No